CLINICAL TRIAL: NCT00965718
Title: Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of Activated T-lymphocyte ("Immuncell-LC") Cell Therapy in Gemcitabine Refractory Advanced Pancreatic Cancer
Brief Title: Evaluate the Efficacy and Safety of Activated T-lymphocyte Cell Therapy in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILC-IIT-01
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Results first posted 2014-09-16 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Cancer
Keywords: advanced pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immuncell-LC group (Experimental): Intravenous dripping of 200 ml (109~2 1010 lymphocytes/60 kg adult) for 1 hour.
  Interventions: Biological: Activated T lymphocyte

INTERVENTIONS:
Biological: Activated T lymphocyte — Intravenous dripping of 200 ml (109~2 1010 lymphocytes/60 kg adult) for 1 hour.
  Other Names: Immuncell-LC

SUMMARY:
Phase 2 Clinical trial to Evaluate the efficacy and safety of activated T-lymphocyte ("Immuncell-LC") cell therapy in Gemcitabine refractory advanced pancreatic cancer

DETAILED DESCRIPTION:
This was designed as a single-center, single group clinical trial, and subjects include patients with pathologically-confirmed Gemcitabine refractory advanced pancreatic cancer.

If subjects agree to participate in the clinical trial by signing a written consent, only appropriate subjects, who meet the criteria on the examinations and tests, will undergo this clinical trial. To participate in the clinical trial, subject's blood of more than 60 ml should be withdrawn to make a study drug at least 2 weeks before administration. Subjects should visit to hospital according to the protocol and receive a study drug. Therapeutic response rate, overall survival rate, time to progression and the quality of life should be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who signed the written consent form by themselves, protectors or legal representatives prior to the clinical trial after the person in charge explained fully about objectives, procedure and the characteristics of the study drug.
2. Patient aged 18 to 75
3. Patient with pathologically-confirmed, advanced pancreatic cancer
4. ECOG scale (ECOG-PS) ≤2 (Appendix 4. Performance status scale/score)
5. Patient with anticipated survival period of more than 3 months
6. Patient with progressed disease after Gemcitabine-based primary anti-cancer chemotherapy
7. Patient whose blood test, renal function test and liver function test results meet the following conditions.

Exclusion Criteria:

1. Patient with the medical history of immunodeficiency or autoimmune disease that could be aggravated by immunotherapy (examples: rheumatoid arthritis, systemic lupus erythematosus, vasculitis, multiple sclerosis, adolescent Insulin-Dependent Diabetes Mellitus, etc.)
2. Confirmed immunodeficient patient
3. Patient with the history of cancer other than skin cancer, local prostate cancer or carcinoma in situ of cervix within the last 5 years of the start of study
4. Patient who has received systemic anti-angiogenic agent
5. Patient who has received a chemotherapy other than Gemcitabine based chemotherapy
6. Obvious myocardial failure or uncontrolled arterial hypertension
7. Patient who has experienced serious allergy (judged by the investigator)
8. Patient with serious psychological disease (judged by the investigator)
9. Pregnant woman, breast-feeding woman or woman who want to be pregnant during the trial period
10. Patient who has participated in another clinical trial within the last 4 weeks of the start of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siyoung Song, MD, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei medical center, Seoul, South Korea

REFERENCES:
- [Derived] Chung MJ, Park JY, Bang S, Park SW, Song SY. Phase II clinical trial of ex vivo-expanded cytokine-induced killer cells therapy in advanced pancreatic cancer. Cancer Immunol Immunother. 2014 Sep;63(9):939-46. doi: 10.1007/s00262-014-1566-3. Epub 2014 Jun 12. PMID 24916038
- See also: Research paper — http://www.ncbi.nlm.nih.gov/pubmed/24916038

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced pancreatic cancer who showed disease progression during gemcitabine-based chemotherapy were enrolled in this study.
  Twenty patients were enrolled between September 2009 and September 2010.
Groups:
- Immuncell-LC Group: Activated T lymphocyte, intravenous dripping of 200ml (10^9~2*10^10 lymphocytes / 60kg adult) for 1 hour.
Period: Overall Study
Arm/Group | Immuncell-LC Group
Started | 20
Completed | 16
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 59.2 [41 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20
ECOG-PS [Number; unit: participants] — Eastern Cooperative Oncology Group performance status (ECOG-PS) is used by researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  "0"-Fully active, able to carry on all pre-disease performance without restriction "1"-Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature "2"-Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  participants
    0 | 12
    1 | 7
    2 | 1
Duration since diagnosis [Median (Full Range); unit: months] | 9.2 [3.8 to 94.6]
Period of prior chemotherapy [Median (Full Range); unit: months] | 5.2 [2.0 to 13.9]
Site of metastasis [Number; unit: participants]
  Liver | 9
  Lung | 6
  Lymph node | 5

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1). Complete Response: Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
  Disease control rate = CR or PR or SD patients / ITT population *100
Time Frame: Every 2 months from the baseline, up to 16 weeks
Population: Patients who underwent response evaluation at least once were included in the intention-to-treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 16
percentage of participants | 25 [3.78 to 46.22]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated from the date of enrollment until death from any cause. And OS was estimated using Kaplan-Meier methods with 95% confidence intervals (CIs).
Time Frame: Every visit, up to 16 weeks
Population: Patients who underwent response evaluation at least once were included in the intention-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 16
weeks | 26.6 [8.6 to 44.6]

3. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: Every 2 months from the baseline, up to 16 weeks
Population: Patients who underwent response evaluation at least once were included in the intention-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 16
weeks | 11 [8.8 to 13.2]

4. Secondary Outcome: Quality of Life (QoL) Assessed Using the Quality of Life Questionnaire Core 30 (QLQ-C30)
Description: QLQ-C30 constitutes a functional scale(physical, role, emotional, cognitive, and social functioning), symptom scores scale(fatigue, nausea/vomiting, pain, dyspnea, constipation, diarrhea, insomnia, appetite loss, financial difficulties), and global QoL scale. With the scores of all scales ranging from 0 to 100, a higher score indicates a better functional scale and a better global QoL scale as well as a worse symptom scores scale.
Time Frame: Every one month from the baseline, up to 16 weeks
Population: Patients who underwent response evaluation at least once were included in the intention-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 16
units on a scale
  Global health status at baseline | 53.65 (29.81) [0.76 to 5.62]
  Global health status at last visit | 40.63 (25.98)
  Physical functioning at baseline | 73.75 (30.64)
  Physical functioning at last visit | 69.58 (21.63)
  Role functioning at baseline | 76.04 (32.76)
  Role functioning at last visit | 59.38 (29.79)
  Emotional functioning at baseline | 70.31 (20.41)
  Emotional functioning at last visit | 61.98 (23.56)
  Cognitive functioning at baseline | 71.88 (24.13)
  Cognitive functioning at last visit | 68.75 (28.46)
  Social functioning at baseline | 68.75 (20.97)
  Social functioning at last visit | 55.21 (27.02)
  Fatigue at baseline | 40.97 (24.59)
  Fatigue at last visit | 50.69 (29.25)
  Nausea/vomiting at baseline | 15.63 (25.44)
  Nausea/vomiting at last visit | 16.67 (18.26)
  Pain at baseline | 20.83 (25.46)
  Pain at last visit | 45.83 (26.87)
  Dyspnea at baseline | 10.42 (20.07)
  Dyspnea at last visit | 27.08 (32.70)
  Constipation at baseline | 16.67 (24.34)
  Constipation at last visit | 29.17 (40.14)
  Diarrhea at baseline | 8.33 (25.82)
  Diarrhea at last visit | 8.33 (19.25)
  Insomnia at baseline | 14.58 (20.97)
  Insomnia at last visit | 43.75 (33.82)
  Appetite loss at baseline | 31.25 (33.26)
  Appetite loss at last visit | 43.75 (37.94)
  Financial difficulties at baseline | 27.08 (30.35)
  Financial difficulties at last visit | 31.25 (33.26)
Statistical Analysis 1: Comparison: Immuncell-LC Group; Test type: Superiority or Other; p = 0.123, t-test, 2 sided — Global health status scores at baseline and final observation point were compared via a 2-sided t-test

5. Secondary Outcome: Quality of Life (QoL) Assessed Using Quality of Life Questionnaire Core 30(QLQ-C30) in Patients With Pancreatic Cancer(QLQ-PAN26 Questionnaire)
Description: QLQ-PAN26 consists of questions (Qs) relating to disease symptoms, treatment (Tx) side effects and emotional issues specific to pancreatic cancer (PC). Questions include on altered bowel habits, pain, dietary changes, disease and Tx-related symptoms and issues related to the emotional and social well-being of participants with PC. All Qs are answered on 4-point Likert scale ranging from '1=not at all' to 4='very much' and subsequently transformed into scales that range from 0-100; higher scores= greater degree of symptoms or treatment side effects and emotional issues.
Time Frame: Every one month from the baseline, up to 16 weeks
Population: Patients who underwent response evaluation at least once were included in the intention-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 16
units on a scale
  Pancreatic pain at baseline | 77.08 (23.07)
  Pancreatic pain at last visit | 60.42 (25.91)
  Gastrointestinal at baseline | 78.13 (29.01)
  Gastrointestinal at last visit | 63.54 (29.32)
  Jaundice at baseline | 93.75 (11.98)
  Jaundice at last visit | 87.50 (16.67)
  Body image at baseline | 56.25 (38.91)
  Body image at last visit | 56.25 (29.74)
  Altered bowel habit at baseline | 79.17 (24.72)
  Altered bowel habit at last visit | 61.46 (24.13)
  Health satisfaction at baseline | 35.42 (24.25)
  Health satisfaction at last visit | 34.38 (27.53)
  Sexuality scale at baseline | 55.21 (39.78)
  Sexuality scale at last visit | 54.17 (34.16)
  Bloated abdomen at baseline | 35.42 (25.73)
  Bloated abdomen at last visit | 54.17 (34.16)
  Taste changes at baseline | 29.17 (29.50)
  Taste changes at last visit | 43.75 (35.94)
  Indigestion at baseline | 27.08 (34.89)
  Indigestion at last visit | 41.67 (31.03)
  Flatulence at baseline | 20.83 (23.96)
  Flatulence at last visit | 33.33 (32.20)
  Weight loss at baseline | 22.92 (33.82)
  Weight loss at last visit | 27.08 (25.00)
  Decreased muscle strength at baseline | 31.25 (30.96)
  Decreased muscle strength at last visit | 43.75 (29.11)
  Dry mouth at baseline | 25.00 (31.03)
  Dry mouth at last visit | 45.83 (34.16)
  Treatment side effects at baseline | 29.17 (36.26)
  Treatment side effects at last visit | 39.58 (30.35)
  Fear for future health at baseline | 52.08 (29.74)
  Fear for future health at last visit | 58.33 (19.25)
  Ability to plan ahead at baseline | 31.25 (33.26)
  Ability to plan ahead at last visit | 52.08 (27.13)
  Average pain at baseline | 1.13 (1.89)
  Average pain at last visit | 3.19 (2.43)

6. Primary Outcome: Stable Disease(SD)
Description: Of the 16 patients in the ITT population, stable disease(SD) was confirmed. Disease control rate was calculated based on the number of CR or PR or SD patients in the ITT population.
Time Frame: Every 2 months from the baseline, up to 16 weeks
Population: Patients who underwent response evaluation at least once were included in the intention-to-treat (ITT) population.
Measure: Number; unit: number of participants
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 16
number of participants | 4

7. Primary Outcome: Progressive Disease(PD)
Description: Of the 16 patients in the ITT population, progressive disease (PD) was confirmed. Disease control rate was calculated based on the number of CR or PR or SD patients in the ITT population.
Time Frame: Every 2 months from the baseline, up to 16 weeks
Population: Patients who underwent response evaluation at least once were included in the intention-to-treat (ITT) population.
Measure: Number; unit: number of participants
Arm/Group | Immuncell-LC Group
Number analyzed (Participants) | 16
number of participants | 12

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were recorded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3.0.
Arm/Group | Immuncell-LC Group
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immuncell-LC Group (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 (2) — Regarded as definitely not related to therapy by investigators.
Ascite (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immuncell-LC Group (N=20)
Vomiting (Gastrointestinal disorders) | 7 (9)
Nausea (Gastrointestinal disorders) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No